CLINICAL TRIAL: NCT03560362
Title: Randomized Trial Comparing Bupivacaine vs Lipossomic Extended Release Bupivacaine for Postoperative Pain Control After Minimally Invasive Thoracic Surgery
Brief Title: Postoperative Pain Control With Lipossomic Extended Release Bupivacaine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Benny Weksler, Professor of Surgery, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-03838
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Pain, Postoperative; Lung Cancer
Keywords: bupivacaine; lipossomal extended release bupivacaine; Intercostal nerve block; thoracic surgery; minimally invasive surgery
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupivacaine with epinephrine (Active Comparator): Patients will receive intraoperative intercostal nerve block with bupivacaine
  Interventions: Drug: Bupivacaine / Epinephrine
- Lipossomal extended release bupivacaine (Experimental): Patients will receive intraoperative intercostal nerve block with lipossomal extended release bupivacaine
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Bupivacaine liposome
  Arms: Lipossomal extended release bupivacaine
Drug: Bupivacaine / Epinephrine
  Arms: Bupivacaine with epinephrine

SUMMARY:
Randomized trial of intraoperative intercostal block with bupivacaine with epinephrine compared to lipossomal extended release bupivacaine.

DETAILED DESCRIPTION:
Patients undergoing minimally invasive thoracic surgery will be randomized to receive 0.05% bupivacaine with 1:200,000 epinephrine (control group) or extended release lipossomal bupivacaine. Primary outcomes are postoperative pain measured by visual analog scale, amount of morphine equivalent narcotics used, and postoperative complications. Patients are excluded if they undergo open thoracotomy, or minimally invasive decortication.

ELIGIBILITY:
Inclusion Criteria: Patients who will be undergoing minimally invasive thoracic surgery

* Patients who will be undergoing minimally invasive thoracic surgery

Exclusion Criteria:

* Open surgery
* Chronic use of narcotics
* Use of pregabalin or similar
* Significant liver or kidney dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07-09 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 3-5 days post op
  Pain assessment with Visual Analog Scale (VAS). This is a numeric pain scale widely used in healthcare that ranks pain from 0 (no pain) to 10 (unbearable pain). A pain score below 3 is considered good.

SECONDARY OUTCOMES:
Postoperative complications | 90 days post op
  Any complication occuring in the first 90 days classified according to the Clavien-Dindo classification.
Narcotic used | 3-5 days post op
  Amount of morphine equivalent dosage used in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Benny Weksler, MD, Principal Investigator — University of Tennessee
Locations (1):
- Methodist University Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No